CLINICAL TRIAL: NCT05252845
Title: A Randomized, Open Label, Single Centre, Phase 2 Trial of the Malaria Vaccine, R21/Matrix-M, to Assess Safety and Immunogenicity of the Vaccine in Thai Adults
Brief Title: Safety and Immunogenicity of the Malaria Vaccine, R21/MatrixM, in Healthy Thai Adults
Acronym: R21/Matrix-M
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAL22001; MR/T006161/1 (Other Grant/Funding Number: Medical Research Council [MRC])
Record Dates: First submitted 2022-01-10; First posted 2022-02-23 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-04

CONDITIONS: Malaria,Falciparum
Keywords: Malaria vaccine; Immunogenicity of the malaria vaccine; Immunologic response to malaria vaccine
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R21/Matrix-M + DHA-PIP+PQ (Experimental): The R21/Matrix-M vaccine (IM injection) + co-formulated Dihydroartemisinin/Piperaquine tablets + one single low dose of Primaquine
  Interventions: Biological: R21/Matrix-M vaccination; Drug: DHA-PIP; Drug: PQ
- R21/Matrix-M only (Experimental): The R21/Matrix-M vaccine (IM injection) only
  Interventions: Biological: R21/Matrix-M vaccination
- DHA-PIP+PQ only (Active Comparator): Co-formulated Dihydroartemisinin/Piperaquine tablets + one single low dose of Primaquine
  Interventions: Drug: DHA-PIP; Drug: PQ

INTERVENTIONS:
Biological: R21/Matrix-M vaccination — R21/Matrix-M is the standard formulation of the vaccine (Once prepared, a standard dose of R21/Matrix-M contains approximately 5 µg of R21 antigen, in 0.5 mL of liquid adjuvant containing 50 µg MatrixM). The reconstituted vaccine will be administered by slow IM injection on Day 0 at Study Months 0, 1 and 2.
  Arms: R21/Matrix-M + DHA-PIP+PQ; R21/Matrix-M only
Drug: DHA-PIP — Dihydroartemisinin/piperaquine tablets for adult patients each contain 40 mg dihydroartemisinin and 320 mg piperaquine with a therapeutic dose range between 2-10 mg/kg/day dihydroartemisinin and 16-26 mg/kg/dose piperaquine. Participants will receive three rounds of antimalarial drugs - each round starting on the day of vaccination (Day 0) at Study Months 0, 1 and 2. Each round consists of three daily doses of co-formulated dihydroartemisinin/piperaquine on Day 0, 1, and 2.
  Arms: DHA-PIP+PQ only; R21/Matrix-M + DHA-PIP+PQ
Drug: PQ — Each participant will receive a single low dose primaquine on the day of vaccination (Day 0) at Month 0, Month 1, and Month 2. One single low dose primaquine of approximately 0.25 mg/kg will be administered.
  Arms: DHA-PIP+PQ only; R21/Matrix-M + DHA-PIP+PQ

SUMMARY:
Malaria remains one of the leading causes of morbidity and mortality worldwide. Plasmodium falciparum is a complex pathogen with numerous immune evasion mechanisms which has added layers of complexity to the development of safe and protective vaccines. There remains an urgent need to identify and develop more protective and more affordable vaccine candidates that could achieve the World Health Organization (WHO) goal of 75% efficacy against clinical malaria.

R21 is a novel pre-erythrocytic candidate malaria vaccine. R21 includes Hepatitis B surface antigen (HBsAg) fused to the C-terminus and central repeats of the circumsporozoite protein of P. falciparum (CSP), which self-assemble into virus-like particles in yeast. R21 lacks the excess HBsAg found and comprises only fusion protein moieties.

R21/MatrixM (MM) had a favourable safety profile and was well tolerated. The majority of adverse events were mild, with the most common event being fever. None of the serious adverse events were attributed to the vaccine. At one year, vaccine efficacy remained high, at 77%. Participants vaccinated with R21/MM showed high titres of malaria-specific anti- Asn-Ala-Asn-Pro (NANP) antibodies 28 days after the third vaccination, which were almost doubled with the higher adjuvant dose. Titres waned but were boosted to levels similar to peak titres after the primary series of vaccinations after a fourth dose administered one year later.

Currently, there are no safety and immunogenicity data for the use of R21/MatrixM in Asian populations. This trial will generate the required data for the use of this vaccine in Asia. For integration with the current targeted malaria elimination (TME) activities, which provide mass drug administrations at months M0, M1, and M2, it would be most efficient and practical to provide the vaccine at the same intervals.

In summary: The investigators propose to conduct a safety and immunogenicity trial of R21/MatrixM in Thai adults. The major aims of this study are to 1) assess the safety and immunogenicity of R21/MatrixM in Thai adults 2) confirm that the co-administration of antimalarial drugs with the malaria vaccine R21/MatrixM does not reduce the immunogenicity of the vaccine and 3) assess the absorption and pharmacokinetics of antimalarial drugs piperaquine, and a single low dose of primaquine (SLDPQ) when co-administered with R21/MatrixM.

This is a randomized, open label, single centre, Phase 2 study. 120 healthy non-pregnant Thai adults, aged 18-55 years, inclusive, will be recruited.

Each participant will be randomized into one of the following study arms in a ratio of 5:5:2, as follows:

1. R21/MatrixM + Dihydroartimisinin (DHA)-Piperaquine (PIP)+ primaquine (PQ) (Group 1, n=50) will receive R21/MatrixM + 3 doses DHA-PIP+PQ at Month 0, Month 1 and Month 2
2. R21/MatrixM only (Group 2, n=50) will receive R21/MatrixM standard dose at Month 0, Month 1 and Month 2
3. DHA-PIP+PQ only (Group 3, n=20) will receive 3 doses DHA-PIP+PQ at Month 0, Month 1 and Month 2

DETAILED DESCRIPTION:
This is a randomized, open label, single centre, Phase 2 study.

Screening and eligibility assessment (Screening visit) All potential volunteers will have a screening visit, which may take place up to 7 days prior to enrolment. Once informed consent is given, a screening number will be assigned in sequential order. Screening numbers will be issued consecutively (e.g. R21-001, R21-002, R21-003, …)

Enrolment, baseline assessment, regimen allocation, and first vaccination (Month 0 / Day 0 visit; Baseline visit) All inclusion and exclusion criteria will be checked before enrolment in the study. Physical examination will be performed. Any new medical issues or symptoms that have arisen will be assessed. Blood will be collected for baseline P. falciparum testing, haemoglobin and biochemistry. Participants with parasitaemia or anaemia will be treated according to national guidelines. Blood will be collected and stored for measurement of antibodies against P. falciparum circumsporozoite (anti-circumsporozoite antibody) until shipment to the reference laboratory. Urine will be collected from women of child-bearing age for immediate pregnancy test.

Enrolment, baseline assessment, regimen allocation, and first vaccination (Month 0 / Day 0 visit; Baseline visit)

All inclusion and exclusion criteria will be checked before enrolment in the study. Physical examination will be performed. Any new medical issues or symptoms that have arisen will be assessed. Blood will be collected for baseline P. falciparum testing, haemoglobin and biochemistry. Blood will be collected and stored for measurement of antibodies against P. falciparum circumsporozoite (anti-circumsporozoite antibody) until shipment to the reference laboratory. Urine will be collected from women of child-bearing age for immediate pregnancy test.

If all inclusion criteria are fulfilled and none of the exclusion criteria apply, the patient will be enrolled into the study and a case record form (CRF) specific to each participant completed. Regimen allocation and administration of the vaccine(s) will be on Day 0. The randomization lists will be prepared by Mahidol-Oxford Tropical Medicine Research Unit (MORU).

Randomization numbers will be generated in blocks, for the 3 study arms in a ratio of 5:5:2, as follows:

* R21/MatrixM + DHA-PIP+PQ (Group 1)
* R21/MatrixM alone (Group 2)
* DHA-PIP+PQ alone (Group 3)

Study participants will be assigned the next available randomization number on the list, and thus will be randomly allocated to Group 1, 2, or 3. This is an open-label study. Participants and clinical investigators will not be blinded to group allocation.

Subjects (in group 1 and 2) will then be vaccinated by intramuscular (IM) needle injection into the deltoid region of the arm. Subjects in Groups 1 and 3 will also receive anti-malarial medications.

The study participants will be observed closely for at least 30 minutes following the administration of each study vaccine, with appropriate medical treatment readily available in case of an anaphylactic reaction.

Subsequent vaccination visits (Month 1 / Day 0 and Month 2 / Day 0 visits)

Physical examination will be performed. Any new medical issues or symptoms that have arisen will be assessed. Blood will be collected for P. falciparum testing. Participants with parasitaemia or anaemia will be treated according to national guidelines. Blood will be collected and stored for measurement of antibodies against P. falciparum circumsporozoite (anti-circumsporozoite) until shipment to the reference laboratory. Urine will be collected from women of child-bearing age for immediate pregnancy test.

Before vaccination, the on-going eligibility of the volunteer will be reviewed. All participants will attend the clinic for vaccination visits, will be observed closely for at least 30 minutes following the administration of each study vaccine.

Follow up assessments

Follow-up assessments (visits not involving vaccination) will be done at month 3 and month 6 after the first vaccination.

Blood tests

Blood will be drawn at the time points indicated in the schedule of procedures and the following laboratory assays performed:

At screening:

* Haematology: haemoglobin (Hb), leukocytes (white blood cells [WBC]) and platelets (PLT).
* Biochemistry: alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine (CREA).
* Diagnostic serology: HBsAg, HCV antibodies, HIV antibodies (Counselling will be given prior to testing blood for these blood-borne viruses)
* P. falciparum testing

At M0, D0: P. falciparum testing, Haematology: Hb, WBC, PLT, Biochemistry: ALT, AST, CREA, anti-circumsporozoite antibody; Pharmacokinetics (piperaquine and primaquine drug levels will be assessed if additional data are required) At M0, D1: Pharmacokinetics (piperaquine and primaquine drug levels) At M0, D2: Pharmacokinetics (piperaquine drug levels) At M0, D7: Haematology: Hb, WBC, PLT; Biochemistry: ALT, AST, CREA; Pharmacokinetics (piperaquine drug levels) At M1, D0: P. falciparum testing, anti-circumsporozoite antibody; Pharmacokinetics (piperaquine drug levels) At M1, D1: Pharmacokinetics (piperaquine and primaquine drug levels) At M1, D2: Pharmacokinetics (piperaquine drug levels) At M1, D7: Haematology: Hb, WBC, PLT; Biochemistry: ALT, AST, CREA; Pharmacokinetics (piperaquine drug levels) At M2, D0: P. falciparum testing, anti-circumsporozoite antibody; Pharmacokinetics (piperaquine drug levels) At M2, D1: Pharmacokinetics (piperaquine and primaquine drug levels) At M2, D2: Pharmacokinetics (piperaquine drug levels) At M2, D7: Haematology: Hb, WBC, PLT; Biochemistry: ALT, AST, CREA; Pharmacokinetics (piperaquine drug levels) At M3: P. falciparum testing, Haematology: Hb, WBC, PLT; Biochemistry: ALT, AST, CREA; anti-circumsporozoite antibody At M6: P. falciparum testing, anti-circumsporozoite antibody

ELIGIBILITY:
Inclusion Criteria

The participant is eligible to enter the study if all of the following apply:

1. Participant is a healthy adult, aged 18 to 55 years (inclusive), of Thai origin.
2. Participant is willing and able to give informed consent to participate in the trial
3. Able, in the investigator's opinion, and willing to comply with the study requirements and follow-up.
4. Women of childbearing potential: must agree to practice continuous, effective contraception for the duration of the trial, and have a negative pregnancy test before each vaccination. (Costs for contraceptives will be reimbursed by the trial.)

Exclusion criteria

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

1. Pregnancy or breastfeeding, or planned pregnancy during the course of the study.
2. Presence of any medical condition (physical or mental) which, may place the participant at undue risk or interfere with the results of the study*. Including: serious cardiac, renal, hepatic or neurological disease, severe malnutrition
3. Any confirmed or suspected immunosuppressive or immunodeficient condition. Including: history of splenectomy, human immunodeficiency virus (HIV) infection
4. Chronic administration (>14 days in total) of immunosuppressants or other immune-modifying drugs within six months of enrollment. Including: oral corticosteroids equivalent to prednisone > 20 mg/day (a)
5. History of an autoimmune disease
6. Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody(b) detected in serum.
7. Screening electrocardiogram (ECG) demonstrating a QTc interval ≥ 450 ms
8. Seropositivity for hepatitis C virus (antibodies to HCV) at screening (b)
9. Finding on safety laboratory values as defined below:

   * AST > 2 x upper normal limit
   * ALT > 2 x upper normal limit
   * Anaemia (Hb < 10 g/dL),
   * Platelets < 150,000
   * Total bilirubin > 2 x upper normal limit
10. Abnormalities of examination or investigations at screening. Including: hepatomegaly, right upper quadrant abdominal pain or tenderness, abnormal blood tests (as defined in the protocol which are not listed above)
11. Positive malaria parasitaemia (RDT) at screening or baseline (Month 0, Day 0).
12. Receipt or planned receipt of an investigational medical product or participation in an interventional clinical trial during the study period
13. Contraindications to the use of artemisinins, piperaquine or primaquine*. Including: use of medications with known potential interactions, prior allergic reactions to one or more components of the drug regimen.
14. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products)
15. History of clinically significant contact dermatitis.
16. Contraindication to intramuscular (IM) injection*
17. Administration of a vaccine not included in the study protocol within 30 days of a study vaccine (c).
18. History of anaphylaxis post-vaccination.
19. Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.

    * subject to the investigator's judgement

Exceptions:

a Inhaled and topical steroids. b Participation in hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study c The following vaccinations may be administered more than 7 days before or after a study vaccination: polio, diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b, Bacillus Calmette-Guérin (BCG vaccine), measles, influenza, pneumococcal disease, COVID-19 or yellow fever

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Hospital for Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All personal details of participants will be de-identified. These data including laboratory investigation results will be stored and may be shared with other researchers to apply in their research in accordance with the MORU data sharing policy.
Time Frame: After completion of trial activities and reporting
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Started | 52 | 53 | 22
Completed | 48 | 48 | 20
Not Completed | 4 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only | Total
Number analyzed (Participants) | 52 | 53 | 22 | 127
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.5 [32 to 45] | 40 [32 to 44] | 40.5 [31.5 to 44] | 40 [32 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 17 | 88
  Male | 19 | 15 | 5 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Median (Inter-Quartile Range); unit: Kg.] | 64.3 [56 to 71.3] | 60.7 [52.1 to 73] | 64 [53.3 to 71.7] | 63.1 [54.1 to 71.7]
the heart rate-corrected QT (QTc) interval [Median (Inter-Quartile Range); unit: Millisecond] | 416 [405 to 426] | 415.5 [401 to 430] | 416 [402 to 429] | 416 [403.5 to 428.5]
Hemoglobin (Hb) [Mean (Standard Deviation); unit: g/dL] | 13.5 (3.9) | 12.9 (1.2) | 12.7 (1.1) | 13.1 (2.6)
White Blood Cell (WBC) [Mean (Inter-Quartile Range); unit: 10^3 cells/Microliter] | 6.4 [5.7 to 7.6] | 7.1 [6.0 to 7.9] | 6.7 [5.3 to 7.9] | 6.5 [5.8 to 7.6]
Platelets [Median (Inter-Quartile Range); unit: 10^6 cells/Microliter] | 281.5 [241 to 307] | 271 [238 to 333] | 262.5 [241 to 310] | 277 [240.5 to 325.5]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.7 [0.7 to 0.9] | 0.7 [0.7 to 0.8] | 0.7 [0.6 to 0.8] | 0.7 [0.7 to 0.9]
Aspartate Aminotransferase (AST) [Median (Inter-Quartile Range); unit: U/L] | 20.5 [17 to 26] | 17.5 [16 to 20] | 19.5 [16.5 to 21.5] | 19 [16 to 22]
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: U/L] | 19 [14 to 26] | 15.5 [12 to 21] | 14 [12.5 to 19] | 17 [13 to 23.5]
Temperature [Mean (Standard Deviation); unit: ºC] | 36.4 (0.4) | 36.4 (0.3) | 36.5 (0.4) | 36.4 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Unsolicited Adverse Events (AEs), According to the Medical Dictionary for Regulatory Activities (MedRA) Classification.
Time Frame: From the date of the first vaccination to 28 days after the last vaccination (up to approximately 1 month)
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 52 | 53 | 22
Participants | 17 | 6 | 4

2. Primary Outcome: Occurrence of Serious Adverse Events (SAEs), According to the MedRA Classification.
Time Frame: During the whole study period, i.e. during a 6-month follow-up period from the receipt of first vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 52 | 53 | 22
Participants | 1 | 0 | 1

3. Primary Outcome: Occurrence of Solicited Adverse Event Within 7 Days of Each Vaccination
Time Frame: Within 7 days of each vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 52 | 53 | 22
Participants | 37 | 36 | 0

4. Secondary Outcome: Number of Participants With Seroconversions in C-Term
Description: Number of Participants with Seroconversions in C-Term
Time Frame: at study Month 1
Measure: Count of Participants; unit: Participants
Groups:
- R21/Matrix-M Only: The R21/Matrix-M vaccine (IM injection)
  R21/Matrix-M vaccination: R21/Matrix-M is the standard formulation of the vaccine (Once prepared, a standard dose of R21/Matrix-M contains approximately 5 µg of R21 antigen, in 0.5 mL of liquid adjuvant containing 50 µg MatrixM). The reconstituted vaccine will be administered by slow IM injection on Day 0 at Study Months 0, 1 and 2.
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 47 | 49 | 18
Participants | 41 | 38 | 0

5. Secondary Outcome: Number of Participants With Seroconversions in C-Term
Description: Number of Participants with Seroconversions in C-Term
Time Frame: at study Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 48 | 19
Participants | 50 | 48 | 3

6. Secondary Outcome: Number of Participants With Seroconversions in C-Term
Description: Number of Participants with Seroconversions in C-Term
Time Frame: at study Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 49 | 48 | 18
Participants | 49 | 48 | 3

7. Secondary Outcome: Number of Participants With Seroconversions in C-Term
Description: Number of Participants with Seroconversions in C-Term
Time Frame: at study Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 48 | 48 | 18
Participants | 48 | 48 | 0

8. Secondary Outcome: Number of Participants With Seroconversions in NANP
Description: Number of Participants with Seroconversions in NANP
Time Frame: at study Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 50 | 20
Participants | 49 | 50 | 1

9. Secondary Outcome: Number of Participants With Seroconversions in NANP
Description: Number of Participants with Seroconversions in NANP
Time Frame: at study Month2
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 50 | 20
Participants | 50 | 49 | 1

10. Secondary Outcome: Number of Participants With Seroconversions in NANP
Description: Number of Participants with Seroconversions in NANP
Time Frame: at study Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 49 | 20
Participants | 50 | 49 | 2

11. Secondary Outcome: Number of Participants With Seroconversions in NANP
Description: Number of Participants with Seroconversions in NANP
Time Frame: at study Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 48 | 48 | 20
Participants | 48 | 48 | 0

12. Secondary Outcome: Number of Participants With Seroconversions in R21
Description: Number of Participants with Seroconversions in R21
Time Frame: at study Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 47 | 50 | 20
Participants | 47 | 50 | 2

13. Secondary Outcome: Number of Participants With Seroconversions in R21
Description: Number of Participants with Seroconversions in R21
Time Frame: at study Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 50 | 20
Participants | 50 | 49 | 3

14. Secondary Outcome: Number of Participants With Seroconversions in R21
Description: Number of Participants with Seroconversions in R21
Time Frame: at study Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 49 | 20
Participants | 50 | 49 | 5

15. Secondary Outcome: Number of Participants With Seroconversions in R21
Description: Number of Participants With Seroconversions in R21
Time Frame: at study Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 48 | 48 | 18
Participants | 48 | 48 | 3

16. Secondary Outcome: Number of Participants With Seroconversions in HBsAg
Description: Number of Participants with Seroconversions in HBsAg
Time Frame: at study Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 49 | 49 | 20
Participants | 27 | 21 | 6

17. Secondary Outcome: Number of Participants With Seroconversions in HBsAg
Description: Number of Participants with Seroconversions in HBsAg
Time Frame: at study Month 2
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 48 | 49 | 20
Participants | 20 | 23 | 2

18. Secondary Outcome: Number of Participants With Seroconversions in HBsAg
Description: Number of Participants with Seroconversions in HBsAg
Time Frame: at study Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 49 | 49 | 20
Participants | 36 | 37 | 4

19. Secondary Outcome: Number of Participants With Seroconversions in HBsAg
Description: Number of Participants with Seroconversions in HBsAg
Time Frame: at study Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
Number analyzed (Participants) | 48 | 48 | 20
Participants | 24 | 26 | 5

20. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (Cmax) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 0
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng/mL | 139 [114 to 185] | 177.5 [125 to 213.5]

21. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (AUC) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 0
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng*h/mL | 23151.6 [19577.8 to 33561.8] | 30594.4 [21015.2 to 36429.7]

22. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (Cmax) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng/mL | 167.0 [116 to 204] | 188.5 [134.5 to 246.0]

23. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (AUC) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 1
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng*h/mL | 24221.4 [16812.2 to 31600.8] | 30672.1 [20366.4 to 38646.6]

24. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (Cmax) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng/mL | 27652 [21772 to 38006.9] | 28055.4 [19286 to 42462.6]

25. Secondary Outcome: For Arms 1 and 3, Piperaquine Levels Following the Administration of the Antimalarials With or Without Vaccine
Description: For Arms 1 and 3, Piperaquine levels (AUC) following the administration of the antimalarials with or without vaccine
Time Frame: Study month 2
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | DHA-PIP+PQ Only
Number analyzed (Participants) | 50 | 20
ng*h/mL | 27652 [21772 to 38006.9] | 28055.4 [19286 to 42462.6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | R21/Matrix-M + DHA-PIP+PQ | R21/Matrix-M Only | DHA-PIP+PQ Only
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/53 | 1/22
Other Adverse Events (participants affected / at risk) | 38/52 | 39/53 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R21/Matrix-M + DHA-PIP+PQ (N=52) | R21/Matrix-M Only (N=53) | DHA-PIP+PQ Only (N=22)
Community-acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis with neuromyelitis optica (NMO) right eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R21/Matrix-M + DHA-PIP+PQ (N=52) | R21/Matrix-M Only (N=53) | DHA-PIP+PQ Only (N=22)
Malaise (General disorders) | 4 (4) | 3 (3) | 0 (0)
Fever (Infections and infestations) | 14 (16) | 9 (9) | 1 (1)
ALT increased (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 14 (18) | 3 (4) | 0 (0)
Somnolence (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Common cold (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Early menstruation (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (General disorders) | 18 (33) | 15 (17) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Community-acquired Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cough (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysplasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eyebrow pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lack of communication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lack of concentration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Left/right jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasm, Ovarian (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash at right little finger (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Running nose (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticarial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sneeze (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (21) | 4 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0)
Fatigue (General disorders) | 21 (42) | 17 (23) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 18 (26) | 23 (29) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 7 (12) | 0 (0)
Chills (General disorders) | 10 (11) | 6 (8) | 0 (0)
Pain (General disorders) | 25 (56) | 30 (56) | 0 (0)
Redness (General disorders) | 3 (6) | 5 (7) | 0 (0)
Swelling (General disorders) | 3 (3) | 10 (12) | 0 (0)
Bruising (General disorders) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT05252845/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT05252845/SAP_001.pdf